CLINICAL TRIAL: NCT02627469
Title: Effect of Weekly Professional Oral Care, During 12 Months, on the Composition of the Oral Flora and Related Variables in Dependent Elderly Residents
Brief Title: Oral Hygiene Care and Microflora in Elderly Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Inger Wårdh, PhD Associate professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KarolinskaII
Record Dates: First submitted 2015-11-04; First posted 2015-12-11 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Pneumonia; Aspiration
Keywords: Microbiota; aged; oral health
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Common oral hygiene help administered by nursing staff
- Intervention (Experimental): Extended professional oral hygiene care Electric toothbrush (Oral-B Professional Care 7000) 1100 ppm sodium fluoride dentifrice (Zendium Classic, Opus Health Care AB/Zendium)
  Interventions: Behavioral: Extended professional oral hygiene care; Device: Electric toothbrush (Oral-B Professional Care 7000); Device: 1100 ppm sodium fluoride dentifrice (Zendium Classic)

INTERVENTIONS:
Behavioral: Extended professional oral hygiene care — Weekly professional oral hygiene performed by dental hygienists
  Arms: Intervention
Device: Electric toothbrush (Oral-B Professional Care 7000) — Weekly professional oral hygiene performed by dental hygienists
  Arms: Intervention
Device: 1100 ppm sodium fluoride dentifrice (Zendium Classic) — Weekly professional oral hygiene performed by dental hygienists
  Arms: Intervention

SUMMARY:
Objective: The effect of weekly professional oral care on the composition of the oral flora in dentate, dependent elderly residents was followed during a 12-month period.

Background: Long-term, regular professional oral hygiene care reduces the total number of microorganisms and oral disease-related microorganisms. Less is known about the effect on the quality/composition of the remaining oral flora.

Materials and methods: Thirty-three subjects were included in the study group and 35 in the control group. Dental status, presence of supragingival-plaque, labial minor gland secretion rate, and prescription medicines were recorded. Microbial samples, collected from supragingival plaque and the dorsum of the tongue, were analyzed using cultivation technique.

DETAILED DESCRIPTION:
Ethics statement The study was approved by the Ethics Committee at the University of Gothenburg, Sweden (Permit Number 039/00).

Study and control groups After giving an informed and written consent to participate, either by the subjects themselves or by a relative or a guardian, 68 subjects were recruited from two nursing homes for elderly persons. The nursing homes, belonging to the same institution and having the same leadership, are situated in the same area of the city. The study group was recruited from one of the nursing homes and consisted of 21 women and 12 men. The control group, recruited from the second nursing home, consisted of 23 women and 12 men. To be included in the study, the subjects had to have at least 10 natural teeth and no removable dentures and be able to follow simple instructions, such as open and close the mouth. The subjects were included in the study in the order they gave their informed consent and fulfilled the inclusion criteria. Throughout the study period, the subjects in both groups were eligible for dental care for dependent individuals, as regulated by law in Sweden, including an oral health care assessment free of charge, basic dental care at subsidized rates, and nursing home personnel trained in oral health care.

Intervention The study group received professional oral care, once a week throughout the 12-month study period, by either of two dental hygienists. The oral care was carried out in the residents´ private rooms with the participant sitting in his/her own chair or lying in bed. The treatment included brushing of the teeth, at labial and lingual sides, with use of an electric toothbrush (Oral-B Professional Care 7000) and a 1100 ppm sodium fluoride dentifrice (Zendium Classic, Opus Health Care AB/Zendium). Inter-dental cleaning was carried out using inter-dental brushes (TePe: TePe, Malmö, Sweden) and toothpicks (TePe Birch: TePe, Malmö, Sweden). Information and training in oral hygiene procedures were given to those in the study group capable to understand instructions.

At the start of the intervention, each subject in the study group, as well as their main responsible nursing aid, received an electric toothbrush of the same kind as was used by the two dental hygienists (Oral-B Professional Care 7000), and instructions and training on how to use the brush. In the control group, the oral health care procedures followed the ordinary routines for the department.

Collection of clinical data and samples for microbial analysis Clinical examinations, measurements of labial minor gland salivary secretion rate, and microbial samplings were performed between 9 and 12 am (by author KL K) and were carried out in the residents´ private rooms. All microbial sampling was performed in duplicate, one week apart. The clinical examination was performed at the first of the two duplicate sampling occasions. Plaque registration followed by the collection of supragingival plaque for microbial analysis was performed at four sites, in that order. The sites selected were interproximally the upper right first and second molars, the lower left first and second molars, the upper right second incisor and the canine, and the lower left second incisor and the canine. If one or more of these teeth were missing, the closest available site was selected. The measurement of the labial minor gland salivary secretion rate, followed by microbial sampling from the tongue, was performed in that order and at the end of the registration and sampling sessions.

In both the study and control groups, clinical data, data on prescription medicines, the labial minor gland salivary secretion rate, and microbial samples were collected at the baseline and at the end of the 12-month study period. In the study group, additional plaque registration and sampling for microbial analysis were performed after 3, 6, and 9 months from the baseline.

Clinical examination The clinical examination was carried out, in the light of an adjustable headlight, using a dental mirror and a dental probe. The number of natural teeth, clinically visible caries lesions and plaque were recorded. Plaque was recorded as no visible plaque (score 0), visible but thin plaque (score 1) or visible thick plaque (score 2). A mean of the plaque scores recorded at the four interproximal sites selected for registration was calculated.

Prescription medicines Data on prescription medicines was collected from the residents´ medical records.

Labial minor gland salivary secretion rate For measurement of the labial minor gland salivary secretion rate, performed as described by Eliasson et al., the area of the lower labial mucosa was gently dried with a cotton pad. A pre-cut piece of a standard filter paper was then placed for 15 s near the midline approximately 3 mm from the outer border of the mucosa. The volume of liquid absorbed by the filter paper was measured using a calibrated Periotron® (8000, ProFlow™ Inc., Amityville, NY, USA). At each examination, four samples were collected from each subject and an individual mean was calculated.

Microbial sampling and analysis Microbial samples were collected from the supragingival plaque and the dorsum of the tongue. An experienced laboratory assistant blinded to which group of subjects, study or control group, and to which of the examination occasions the samples were collected from, analyzed the samples.

The supragingival plaque samples were collected using sterile toothpicks (TePe Birch) and pooled. The tongue samples were collected using sterile tweezers, cotton pellets and plastic spatulas. The spatula, with a circular hole 1.5 cm diameter, was placed on the back part of the dorsum. A cotton pellet, immersed in sampling fluid, was swept over the area inside the hole. The two samples were each transferred to 3.5 ml of transport medium VMGA III and processed within four hours.

The analyses of the samples were performed as previously described using enriched blood agar plates and selective agar plates. The total number of microorganisms growing under anaerobic conditions, the total number and proportion of streptococci and the number and proportion of Streptococcus sanguinis/oralis and Streptococcus salivarius, both associated with good oral health, mutans streptococci, lactobacilli and Actinomyces spp, associated with dental caries, F. nucleatum, and P. intermedia/nigrescens, associated with gingival inflammation, P. gingivalis and A. actinomycetemcomitans, associated with periodontitis, Candida albicans, Staphylococcus aureus, and enteric rods, associated with mucosal and aspiratory infections, were calculated. The detection limit was 100 colony-forming units for all species except A. actinomycetemcomitans, where the detection limit was 10 colony-forming units. If possible, the number of microorganisms was calculated from their number on a plate giving 30 - 300 colonies. A mean of the results from the duplicate samplings was calculated.

Statistical methods To normalize the microbial data, the numbers were transformed logarithmically. Zero counts were treated as one colony forming unit/ml. Mean and median values and standard deviations were calculated. One-way ANOVA was used for the analysis of differences between the study and control groups. Two-way ANOVA was used for statistical analysis of differences at different time points within the two groups. Results were regarded statistically significant at p-values < 0.05. Owing to the multiple influence aspect, isolated significances should be interpreted with some caution.

ELIGIBILITY:
Inclusion criteria

* 10 or more natural teeth
* no removable dentures
* no or mild cognitive impairments

Exclusion criteria

* less than 10 natural teeth
* removable dentures
* severe cognitive impairments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Composition of the oral microflora | 12 months
  Microbial samples were collected from the supragingival plaque and the dorsum of the tongue.
  The total number of microorganisms growing under anaerobic conditions, the total number and proportion of streptococci, lactobacilli, Actinomyces spp, F. nucleatum, P. intermedia/nigrescens, P. gingivalis, A. actinomycetemcomitans, Candida albicans, Staphylococcus aureus, and enteric rods, were calculated.
  The detection limit was 100 colony-forming units for all species except A. actinomycetemcomitans, where the detection limit was 10 colony-forming units. If possible, the number of microorganisms was calculated from their number on a plate giving 30 - 300 colonies. A mean of the results from the duplicate samplings was calculated.

SECONDARY OUTCOMES:
Rate of Labial minor gland salivary secretion | 12 months
  For measurement of the labial minor gland salivary secretion rate, the area of the lower labial mucosa was gently dried with a cotton pad. A pre-cut piece of a standard filter paper was then placed for 15 s near the midline approximately 3 mm from the outer border of the mucosa. The volume of liquid absorbed by the filter paper was measured using a calibrated Periotron® (8000, ProFlow™ Inc., Amityville, NY, USA). At each examination, four samples were collected from each subject and an individual mean was calculated.
Presence of supragingival-plaque | 12 months
  Plaque was recorded as no visible plaque (score 0), visible but thin plaque (score 1) or visible thick plaque (score 2). A mean of the plaque scores recorded at the four interproximal sites selected for registration was calculated.
Dental status | 12 month
  A clinical examination was carried out, in the light of an adjustable headlight, using a dental mirror and a dental probe. The number of natural teeth and clinically visible caries lesions were recorded.

OTHER OUTCOMES:
Prescription medicines | 12 months
  Data on prescription medicines was collected from the residents´ medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Wårdh, Assoc prof, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Yes
Published data will not be able to connect with an specific individual but each participant is allowed to by request take part of their own data.
Time Frame: 20180810
Access Criteria: Public

REFERENCES:
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov/pubmed?otool=karolib — The study is reported in the paper: Effect of 12-month weekly professional oral hygiene care on the composition of the oral flora in dentate, dependent elderly residents: A prospective study. Wikström M, Kareem KL, Almståhl A, Palmgren E, Lingström P, Wårdh I. Gerodontology. 2017 Jun;34(2):240-248